CLINICAL TRIAL: NCT01426854
Title: Clinical Evaluation of Safety and Efficacy of Nepafenac Ophthalmic Suspension, 0.1% Compared to Placebo for the Prevention and Treatment of Ocular Inflammation and Pain Associated With Cataract Surgery in Adult Chinese Subjects
Brief Title: Nepafenac Compared to Placebo for Ocular Pain and Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-10-026
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Cataract
Keywords: Cataract Surgery; Anti-ocular Inflammation; Anti-ocular Pain
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nepafenac (Active Comparator): Nepafenac Ophthalmic Suspension, 0.1%, 1 drop to the operative eye, 3 times a day, beginning 1 day preoperatively and continuing through the day of surgery and for 14 days postoperatively. An additional dose was administered prior to surgery.
  Interventions: Drug: Nepafenac Ophthalmic Suspension, 0.1%
- Placebo (Placebo Comparator): Nepafenac Vehicle, 1 drop to the operative eye, 3 times a day, beginning 1 day preoperatively and continuing through the day of surgery and for 14 days postoperatively. An additional dose was administered prior to surgery.
  Interventions: Other: Nepafenac Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Nepafenac Ophthalmic Suspension, 0.1% — Topical ocular administration
  Arms: Nepafenac
Other: Nepafenac Vehicle Ophthalmic Solution — Inactive ingredients used as placebo; topical ocular administration
  Arms: Placebo

SUMMARY:
The purpose of this study was to demonstrate that Nepafenac Ophthalmic Suspension, 0.1% is superior to Nepafenac Vehicle (placebo) for the prevention and treatment of ocular inflammation and pain associated with cataract surgery in Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese subjects, 18 years of age or older, of either sex who have a cataract, and are expected to undergo cataract extraction with the implantation of a posterior chamber intraocular lens;
* Study eye of subjects, who in the opinion of the Investigator, will have improvement in best-corrected visual acuity after surgery;
* Subjects should be able to understand and sign an informed consent that has been approved by an Independent Ethics Committee;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Use of topical ocular or systemic steroids within 14 days prior to surgery;
* Use of topical ocular or systemic non-steroidal anti-inflammatory drugs within 7 days of surgery, except an allowed daily dose of baby aspirin (81 mg);
* Subjects planning to have cataract surgery in their fellow, non-study eye prior to the 14 day postoperative study visit;
* Any intraocular inflammation or ocular pain greater than Grade 0 in the study eye that is present during the baseline slit-lamp exam;
* Women of childbearing potential (those who are not surgically sterilized or post menopausal) may not participate in the study if any of the following conditions exist:

  * they are breast feeding;
  * they have a positive urine pregnancy test at baseline;
  * they are not willing to undergo a urine pregnancy test upon exiting the study;
  * they intend to become pregnant during the duration of the study; or,
  * they do not agree to using adequate birth control methods for the duration of the study.
* Any abnormality that prevents reliable tonometry;
* Planned multiple procedures during cataract/IOL implantation surgery;
* Lens pseudoexfoliation syndrome with glaucoma or zonular compromise;
* Previous ocular trauma to the operative eye;
* A history of chronic or recurrent inflammatory eye disease;
* Ocular infection or ocular pain;
* Proliferative diabetic retinopathy;
* Uncontrolled diabetes mellitus;
* Congenital ocular anomaly;
* Iris atrophy in the operative eye;
* A nonfunctional fellow eye;
* Use of an investigational intraocular lens;
* Participation in any other clinical study within 30 days before surgery;
* Known or suspected allergy or hypersensitivity to non-steroidal anti-inflammatory agents, or to any component of the study medication;
* Subjects with known bleeding tendencies, or who are receiving medications that may prolong bleeding time, may be enrolled at the physician's discretion; continuation of previous therapy for these subjects will be left to the judgment of the physician;
* The fellow eye of an individual currently or previously enrolled in the study;
* Subjects using a topical ophthalmic prostaglandin;
* Subjects, who in the opinion of the investigator, might be at increased risk of complications from topical NSAIDs;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Ye, Director, Study Director — Alcon (China) Ophthalmic Product Co., Ltd.
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 study centers in China. Chinese men or women of at least 18 years of age who needed cataract extraction with implantation of a posterior chamber intraocular lens were enrolled and randomized in a ratio of 1:1 to receive either nepafenac or placebo.
Pre-assignment Details: This reporting group includes all enrolled participants.
Period: Overall Study
Arm/Group | Nepafenac | Placebo
Started | 131 | 129
Completed | 119 | 98
Not Completed | 12 | 31
Not completed — Adverse Event | 1 | 5
Not completed — Subject Decision Unrelated to AE | 5 | 6
Not completed — Lost to Follow-up | 3 | 0
Not completed — Noncompliance | 0 | 1
Not completed — Treatment Failure | 0 | 16
Not completed — Protocol Deviation | 0 | 1
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Population: Demographics are presented for the 248 participants who received at least one dose of study drug or discontinued before surgery and failed to return the test article bottle or returned the bottle with a broken seal.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nepafenac | Placebo | Total
Number analyzed (Participants) | 125 | 123 | 248
Age Continuous [Mean (Standard Deviation); unit: years] | 68.8 (10.62) | 69.8 (10.19) | 69.3 (10.40)
Age, Customized [Number; unit: participants]
  18 to <65 years | 35 | 33 | 68
  65 to <75 years | 43 | 44 | 87
  75 to <85 years | 42 | 43 | 85
  85 to <95 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 72 | 144
  Male | 53 | 51 | 104
Region of Enrollment [Number; unit: participants]
  China | 125 | 123 | 248

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Clinical Cure at Day 14
Description: Ocular inflammation was assessed by the Investigator during slit lamp examination. Aqueous cells were scored on a 5-unit scale from 0 (none) to 4 (>30 cells), and aqueous flare (protein escaping from dilated vessels) was scored on a 4-unit scale from 0 (no visible flare when compared with the normal eye) to 3 (severe - very dense flare). To be considered cured, the patient must have had a score of 0 for both aqueous cells and aqueous flare. The proportion of subjects with a clinical cure is reported as percentage.
Time Frame: Day 14 postoperative
Population: Intent-to-treat: All randomized subjects who completed cataract/IOL implant surgery and returned for at least one postoperative primary efficacy assessment.
Measure: Number; unit: Percentage of subjects
Arm/Group | Nepafenac | Placebo
Number analyzed (Participants) | 122 | 122
Percentage of subjects | 80.3 | 39.3
Statistical Analysis 1: Comparison: Nepafenac vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Proportion of Subjects Who Were Pain-Free at All Postoperative Visits
Description: Ocular pain is defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching. The Investigator scored ocular pain based on the description of pain by the subject. Pain was scored on a 6-unit scale ranging from 0 (none, absence of positive sensation) to 5 (severe, subject reports intense ocular, periocular or radiating pain requiring prescription analgesic). To be considered pain-free at all post operative visits, the patient must have had a score of 0 at Days 1, 3, 7, and 14 and any unscheduled visit. The proportion of subjects who were pain-free at all post-operative visits is reported as percentage.
Time Frame: Up to Day 14
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Nepafenac | Placebo
Number analyzed (Participants) | 122 | 122
Percentage of subjects | 71.3 | 40.2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. Individual adverse events were recorded from the start of study treatment. At each visit, after the subject spontaneously mentioned any problems, the study staff inquired about adverse events.
Description: The safety population includes all participants who received at least one dose of study drug or discontinued before surgery and failed to return the test article bottle or returned the bottle with a broken seal.
Arm/Group | Nepafenac | Placebo
Serious Adverse Events (participants affected / at risk) | 0/125 | 1/123
Other Adverse Events (participants affected / at risk) | 0/125 | 0/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nepafenac (N=125) | Placebo (N=123)
Vascular headache (Nervous system disorders) | 0 | 1 — Not related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results, materials of research, relevant intellectual property, and trial materials may not be used, disclosed, revealed, or published in any form without Sponsor's prior written consent.